CLINICAL TRIAL: NCT03748641
Title: A Phase 3 Randomized, Placebo-controlled, Double-blind Study of Niraparib in Combination With Abiraterone Acetate and Prednisone Versus Abiraterone Acetate and Prednisone in Subjects With Metastatic Prostate Cancer
Brief Title: A Study of Niraparib in Combination With Abiraterone Acetate and Prednisone Versus Abiraterone Acetate and Prednisone for Treatment of Participants With Metastatic Prostate Cancer
Acronym: MAGNITUDE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108534; 64091742PCR3001 (Other: Janssen Research & Development, LLC); 2017-003364-12 (EudraCT Number); 2023-503254-12-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Castration-Resistant Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — niraparib; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Participants with mCRPC and HRR Gene Alteration (Experimental): Participants with L1 metastatic castration-resistant prostate cancer (mCRPC) and homologous recombination repair (HRR) gene alteration will receive combination of niraparib 200 milligrams (mg) or matching placebo and abiraterone acetate (AA) 1000 mg plus prednisone 10 mg. In the open label extension (OLE) phase participants earlier receiving the combination of niraparib and AAP may continue to receive open-label combination of niraparib 200 mg and AA 1000 mg plus prednisone 10 mg and those receiving placebo and AAP may cross over depending on the outcome of study to receive open-label combination of niraparib 200 mg and AA 1000 mg plus prednisone 10 mg.
  Interventions: Drug: Niraparib; Drug: Abiraterone Acetate; Drug: Prednisone; Drug: Placebo
- Cohort 2: Participants with mCRPC and No HRR Gene Alteration (Experimental): Participants with L1 mCRPC and no HRR Gene alteration will receive combination of niraparib 200 mg or matching placebo and AA 1000 mg plus prednisone 10 mg. In the OLE phase participants earlier receiving the combination of niraparib and AAP may continue to receive open-label combination of niraparib 200 mg and AA 1000 mg plus prednisone 10 mg and those receiving placebo and AAP may cross over depending on the outcome of study to receive open-label combination of niraparib 200 mg and AA 1000 mg plus prednisone 10 mg.
  Interventions: Drug: Niraparib; Drug: Abiraterone Acetate; Drug: Prednisone; Drug: Placebo
- Cohort 3 (Open-label): Participants with mCRPC (Experimental): Participants with mCRPC will receive a new formulation of niraparib 200 mg and AA 1000 mg tablets plus prednisone 10 mg.
  Interventions: Drug: Prednisone; Drug: New Formulation of Niraparib and Abiraterone Acetate (AA)

INTERVENTIONS:
Drug: Niraparib — Participants will receive niraparib 200 mg capsules or tablets once daily.
  Other Names: JNJ-64091742
  Arms: Cohort 1: Participants with mCRPC and HRR Gene Alteration; Cohort 2: Participants with mCRPC and No HRR Gene Alteration
Drug: Abiraterone Acetate — Participants will receive AA 1000 mg tablets once daily.
  Arms: Cohort 1: Participants with mCRPC and HRR Gene Alteration; Cohort 2: Participants with mCRPC and No HRR Gene Alteration
Drug: Prednisone — Participants will receive prednisone 10 mg tablets daily.
Drug: Placebo — Participants will receive matching placebo once daily.
  Arms: Cohort 1: Participants with mCRPC and HRR Gene Alteration; Cohort 2: Participants with mCRPC and No HRR Gene Alteration
Drug: New Formulation of Niraparib and Abiraterone Acetate (AA) — Participants will receive a new formulation of niraparib 200 mg and AA 1000 mg tablets once daily.
  Arms: Cohort 3 (Open-label): Participants with mCRPC

SUMMARY:
The purpose of this study is to evaluate the effectiveness of niraparib in combination with abiraterone acetate plus prednisone (AAP) compared to AAP and placebo.

ELIGIBILITY:
Inclusion Criteria:

* HRR gene alteration (as identified by the sponsor's required assays) as follows:

  1. Cohort 1: positive for HRR gene alteration
  2. Cohort 2: not positive for DRD (that is, HRR gene alteration)
  3. Cohort 3: eligible by HRR status
* Metastatic disease documented by positive bone scan or metastatic lesions on computed tomography (CT) or magnetic resonance imaging (MRI)
* Metastatic prostate cancer in the setting of castrate levels of testosterone less than or equal to (<=) 50 nanogram per deciliter (ng/dL) on a gonadotropin releasing hormone analog (GnRHa) or bilateral orchiectomy
* Able to continue GnRHa during the study if not surgically castrate
* Score of <= 3 on the brief pain inventory-short form (BPI-SF) question number 3 (worst pain in last 24 hours)

Exclusion Criteria:

* Prior treatment with a poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor
* Systemic therapy (that is, novel second-generation AR-targeted therapy such as enzalutamide, apalutamide, or darolutamide; taxane-based chemotherapy, or more than 4 months of abiraterone acetate plus prednisone [AAP] prior to randomization) in the metastatic castration-resistant prostate cancer (mCRPC) setting; or AAP outside of the mCRPC setting
* Symptomatic brain metastases
* History or current diagnosis of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Other prior malignancy (exceptions: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission) <= 2 years prior to randomization, or malignancy that currently requires active systemic therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2027-02-27 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (317):
- United States (47):
  - Urology Centers Of Alabama, Homewood, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Urological Associates of Southern Arizona, P.C., Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Kaiser Permanente, Riverside, California
  - San Bernardino Urological Associates, San Bernardino, California
  - University of California San Francisco, San Francisco, California
  - Sansum Clinic Pharm, Santa Barbara, California
  - The Urology Center of Colorado, Denver, Colorado
  - Colorado Clinical Research, Lakewood, Colorado
  - VA Connecticut Healthcare, West Haven, Connecticut
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Advanced Urology Institute, Daytona Beach, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Division Of Hematology/oncology, Jacksonville, Florida
  - Veterans Affairs Medical Ctr, Hines, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - First Urology, Jeffersonville, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Healthcare, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Rcca Md, Llc, Bethesda, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Massachusetts General, Boston, Massachusetts
  - Michigan Institute of Urology, Troy, Michigan
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Adult Pediatric Urology & Urogynecology, P.C, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Delaware Valley Urology, LLC, Mount Laurel, New Jersey
  - New York Oncology Hematology, Albany, New York
  - Icahn School of Medicine at Mount Sinai - The Derald H. Ruttenberg, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Upstate Cancer Center, Syracuse, New York
  - Helios Clinical Research, LLC, Middleburg Heights, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Lancaster Urology, Lancaster, Pennsylvania
  - VA Pittsburgh, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Houston Metro Urology, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Salem VA Medical Center, Salem, Virginia
  - Urology of Virginia, PLCC, Virginia Beach, Virginia
  - NorthWest Medical Specialties, PLLC, Tacoma, Washington
- Argentina (12):
  - Hospital Aleman, Buenos Aires
  - Centro Oncológico Korben, Buenos Aires
  - CEMIC Saavedra, Buenos Aires
  - Centro de Urologia (CDU), Ciudad Automoma Buenos Aires
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
  - Hospital Privado de Comunidad, Mar del Plata
  - Centro de Investigacion Pergamino SA, Pergamino
  - Sanatorio Britanico de Rosario, Rosario
  - Sanatorio Parque, Rosario
  - ARS Médica, San Salvador de Jujuy
- Australia (14):
  - Royal Adelaide Hospital, Adelaide
  - Pindara Private Hospital, Benowa
  - Sunshine Coast University Hospital, Birtinya
  - Princess Alexandra Hospital, Brisbane
  - St Vincent s Hospital Sydney, Darlinghurst
  - Royal Hobart Hospital, Hobart
  - Macquarie University, Macquarie University
  - Eye Surgery Associates, Malvern
  - Peter MacCallum Cancer Centre, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Hollywood Private Hospital, Nedlands
  - Prince Of Wales Hospital, Randwick
  - Sydney Adventist Hospital, Wahroonga
  - Wollongong Private Hospital, Wollongong
- Belgium (6):
  - OLV Ziekenhuis Aalst, Aalst
  - ZAS Augustinus, Antwerp
  - Grand Hopital de Charleroi, site Notre Dame, Charleroi
  - AZ Maria Middelares, Ghent
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
  - ZNA Jan Palfijn, Merksem
- Brazil (29):
  - Fundacao Pio XII, Barretos
  - PERSONAL Oncologia de Precisao e Personalizada, Belo Horizonte
  - Sociedade Beneficente de Senhoras - Hospital Sirio Libanes HSL Unidade Brasilia, Brasília
  - CIONC Centro Integrado de Oncologia de Curitiba, Curitiba
  - Pronutrir, Fortaleza
  - Associacao de Combate ao Cancer em Goias - Hospital de Cancer Araujo Jorge, Goiânia
  - Oncosite - Centro de Pesquisa Clínica em Oncologia Ltda, Ijuí
  - Fundacao Sao Francisco Xavier, Ipatinga
  - Instituto Joinvilense de Hematologia e Oncologia Ltda Centro de Hematologia e Oncologia, Joinville
  - Medradius Clinica de Medicina Nuclear e Radiologia de Maceio Ltda., Maceió
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Universidade do Estado do Rio de Janeiro - UERJ, Rio de Janeiro
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Hospital Santa Isabel, Salvador
  - Fundacao do ABC Centro Universitario FMABC, Santo André
  - Irmandade Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
  - Fundacao Faculdade de Medicina Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual IAMSPE, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
  - IOS - Instituto de Oncologia de Sorocaba Dr. Gilson Delgado, Sorocaba
  - Instituto do Cancer De Tres Lagoas, Três Lagoas
- Bulgaria (6):
  - MHAT Deva Maria, Burgas
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - Specialized Hospital for Active Treatment in Oncology EAD, Sofia
  - SHATOD 'Dr. Marko Antonov Markov', Varna
  - Comprehensive Cancer Center, Vratsa
- Canada (9):
  - Southern Alberta Institute of Urology / Prostate Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency BCCA Vancouver Centre, Vancouver, British Columbia
  - British Columbia Cancer Agency Vancouver Island Centre, Victoria, British Columbia
  - McMaster Institute of Urology, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario (Kingston Regional Cancer Centre), Kingston, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - Centre de Recherche du CHUM, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- China (26):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing Cancer Hospital of Peking University, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Hospital, Beijing
  - Sichuan Provincial Peoples Hospital, Chengdu
  - Southwest Hospital, The Third Military Medical University, Chongqing
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat-Sen Memorial Hospital Sun Yat-sen University, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Drug clinical trial ethics committee of Ningbo First Hospital, Ningbo
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Huashan Hospital Fudan University, Shanghai
  - ShangHai Huadong Hospital, Shanghai
  - The Fifth People's Hospital of Shanghai, Fudan University, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Hospital, Tianjin
  - The Central Hospital of Wuhan, Wuhan
  - Tongji Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Wuxi People s Hospital, Wuxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- Czechia (8):
  - Fakultni nemocnice Hradec Kralove, Hradec Králove
  - Krajská nemocnice Liberec, Liberec
  - Uromedical Center s.r.o., Olomouc
  - Multiscan s.r.o., Pardubice
  - Fakultni nemocnice Plzen, Urologicka klinika, Pilsen
  - Urologicka klinika 1 LF UK a VFN, Prague
  - Thomayerova nemocnice, Onkologicka klinika, Prague
  - Uherskohradistska nemocnice a.s., Uherské Hradiště
- France (11):
  - CHRU De Besancon, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Institut Regional du Cancer de Montpellier Val d'Aurelle, Montpellier
  - Polyclinique de Gentilly, Nancy
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges-Pompidou, Paris
  - Institut de Cancerologie de l Ouest ICO, Saint-Herblain
  - HIA Begin, Saint-Mandé
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
- Germany (6):
  - Städtisches Klinikum Braunschweig gGmbH - Standort Salzdahlumer, Braunschweig
  - Urologicum Duisburg, Duisburg
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Universitaetsklinikum Muenster, Münster
  - Studienpraxis Urologie Drs. Feyerabend, Nürtingen
- Hungary (8):
  - Semmelweis Egyetem, Urológia Klinika, Budapest
  - Országos Onkológiai Intézet, C Belgyógyászati-Onkológiai és Klinikai Farmakológiai Osztály, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Josa Andras Oktatokorhaz, Nyíregyháza
  - Uro-Clin Kft., Pécs
  - Szegedi Tudomanyegyetem, Szeged
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- Israel (4):
  - Asaf Harofe Medical Center, Beer Yaakov
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center Tel Hashomer, Ramat Gan
- Italy (13):
  - AUSL Romagna - Ospedale di Faenza, Faenza
  - Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Oncologia Medica A - Ist Naz Tumori G Pascale, Napoli
  - Istituto Oncologico Veneto Iov Irccs Padova, Padua
  - Oncologia Medica - Azienda Ospedaliero Universitaria Di Parma, Parma
  - Ospedale S. Maria Della Misericordia Centro Operativo Studi Clinici SC Oncologia Medica, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - Campus Bio Medico di Roma, Roma
  - Azienda Ospedaliera S. Maria Terni, Terni
  - A.O.U. Città della Salute e della Scienza, Torino
  - Ospedale Santa Chiara Trento, Trento
- Malaysia (6):
  - Hospital Pulau Pinang, George Town
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Likas, Kota Kinabalu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Mexico (5):
  - iBiomed Research Unit, Aguascalientes
  - Consultorio de Especialidad en Urologia Privado, Durango
  - Mexico Centre for Clinical Research, S.A. de C.V., Mexico City
  - Avix Investigacion Clinica S C, Monterrey
  - Consultorio Privado, Zapopan
- Netherlands (7):
  - Antoni van Leeuwenhoek, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - MC Haaglanden Lok Antoniushove - Afd.Interne - INT, Leidschendam
  - St. Antonius Ziekenhuis (St. Antonius Hospital), Nieuwegein
  - Canisius-Wilhelminaziekenhuis, Nijmegen
  - Erasmus MC, Rotterdam
  - Zuyderland Medical Center, Sittard-Geleen
- Poland (9):
  - Szpital Uniwersytecki NR 1 IM Dr Antoniego Jurasza, Bydgoszcz
  - Centrum Onkologii im Prof F Lukaszczyka, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpitale Pomorskie Sp z o o, Gdynia
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Urologica Praktyka Lekarska Adam Marcheluk, Siedlce
  - Pomorski Uniwersytet Medyczny w Szczecinie, Szczecin
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
  - Dolnoslaskie Centrum Onkologii, Wroclaw
- Portugal (5):
  - Hospitais da universidade de Coimbra, Coimbra
  - Instituto Portugues de Oncologia de Coimbra Francisco Gentil, EPE, Coimbra
  - Champalimaud Foundation Champalimaud Centre, Lisbon
  - Centro Hospitalar Lisboa Norte EPE Hosp. Santa Maria, Lisbon
  - H. Santo António - Centro Hospitalar do Porto, Porto
- VA Caribbean Healthcare System, San Juan, Puerto Rico
- Russia (18):
  - Altai Regional Oncology Dispensary, Barnaul
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - GUZ Kursk Regional Oncology Dispensary, Kursk
  - Russian Scientific Center of Roentgenoradiology, Moscow
  - Moscow City Clinical Hospital # 62, Moscow
  - Clinical Diagnostic Centre of Nizhny Novgorod Region, Nizhny Novgorod
  - Clinical Oncology Dispensary, Omsk
  - LLC Novaya Clinica, Pyatigorsk
  - Pyatigorsk Interdistrict Oncology Dispensary, Pyatigorsk
  - Leningrad Regional Oncology Dispensary, Saint Petersburg
  - Private Medical Institution Euromedservice, Saint Petersburg
  - Russian Scientific Center of Radiology and Surgical Technologies, Saint Petersburg
  - Republican Oncology Dispensary, Saransk
  - Oncologic Dispensary No.2, Sochi
  - Tambov Regional Oncology Clinical Dispansary, Tambov
  - Tomsk Cancer Research Institute, Tomsk
  - Medical-sanitary unit 'Neftyanik', Tyumen
  - Vologda Regional Oncological Dispensary, Vologda
- South Africa (2):
  - Clinresco Centres Pty Ltd, Johannesburg
  - Clinical Research Unit, Pretoria
- South Korea (14):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - National Cancer Center, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (12):
  - Hospital Juan Canalejo, A Coruña
  - Hosp. Del Mar, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Univ. I Politecni La Fe, Valencia
- Sweden (3):
  - Sodersjukhuset, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Taiwan (8):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Tungs' Taichung MetroHarbor Hospital, Taichung
  - Chi Mei Medical Center Yong Kang, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (10):
  - Cukurova University, Faculty of Medicine, Adana
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Bakirkoy Training and Research Hospital, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - IEU Medical Point Hospital, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
- Ukraine (12):
  - CNE Clinical Center of Oncology Hematology Transplantology and Palliative Care of the Cherkasy RC, Cherkasy
  - Ce 'Dnipropetrovsk Regional Clinical Hospital N.A. Mechnikov' of Dnipropetrovsk Rc, Dnipo
  - Municipal Institution 'Clinical Oncology Dispensary' Under Dnipropetrovsk Regional Council, Dnipro
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk City Multifield Clinical Hospital # 4, Dnipro
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Municipal non-profit enterprise 'Regional Center of Oncology', Khakhiv
  - Regional Clinical Center of Urology and Nephrology n.a. V.I. Shapoval, Kharkiv
  - State Nonprofit Enterprise National Cancer Institute, Kyiv
  - State Institution Institute of Urology NAMS of Ukraine based on Kyiv City Clinical Oncology Center, Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Council 'Lviv Regional Clinical Hospital', Lviv
  - ME 'Poltava Regional Clinical Hospital n.a. M.V. Sklifosovsky of the Poltava Regional Council', Poltava
  - Municipal Oncology Centre of Uzhgorod Central Municipal Clinical Hospitlal, Uzhhorod
- United Kingdom (6):
  - Royal Blackburn Hospital, Blackburn
  - Royal Lancaster Infirmary, Lancaster
  - UCL Cancer Institute, London
  - Torbay Hospital-Devon, Torquay
  - Royal Cornwall Hospitals NHS Trust - Royal Cornwall Hospital, Truro
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Rathkopf DE, Roubaud G, Chi KN, Efstathiou E, Attard G, Olmos D, Small EJ, Saad M, Castro E, Kim W, Wu D, Bertzos K, Dibaj S, Zhang J, Francis P, Smith MR. Patient-reported Outcomes for Patients with Metastatic Castration-resistant Prostate Cancer and BRCA1/2 Gene Alterations: Final Analysis from the Randomized Phase 3 MAGNITUDE Trial. Eur Urol. 2025 Oct;88(4):359-369. doi: 10.1016/j.eururo.2024.09.003. Epub 2024 Sep 23. PMID 39317633
- [Derived] Roubaud G, Attard G, Boegemann M, Olmos D, Trevisan M, Antoni L, Pascoe K, Capone C, Van Sanden S, Hashim M, Palmer S, Chi K. Adjustment for imbalances in baseline characteristics in the MAGNITUDE phase 3 study confirms the clinical benefit of niraparib in combination with abiraterone acetate plus prednisone in patients with metastatic prostate cancer. Eur J Cancer. 2024 Sep;209:114183. doi: 10.1016/j.ejca.2024.114183. Epub 2024 Jun 17. PMID 39111209
- [Derived] Chi KN, Rathkopf D, Smith MR, Efstathiou E, Attard G, Olmos D, Lee JY, Small EJ, Pereira de Santana Gomes AJ, Roubaud G, Saad M, Zurawski B, Sakalo V, Mason GE, Francis P, Wang G, Wu D, Diorio B, Lopez-Gitlitz A, Sandhu S; MAGNITUDE Principal Investigators. Niraparib and Abiraterone Acetate for Metastatic Castration-Resistant Prostate Cancer. J Clin Oncol. 2023 Jun 20;41(18):3339-3351. doi: 10.1200/JCO.22.01649. Epub 2023 Mar 23. PMID 36952634

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg: Participants with metastatic castration-resistant prostate cancer (mCRPC) and positive homologous recombination repair (HRR) gene alteration, received niraparib 200 milligrams (mg) capsule in combination with abiraterone acetate 1000 mg tablet orally once daily (QD) and prednisone 5 mg tablet orally twice daily (BID) (total dose 10 mg) in each 28 days treatment cycle starting from Cycle 1 Day 1 up to 29 months. Participants were then followed up for safety up to 5 years after last dose or until death, loss to follow-up, withdrawal of consent, or study termination. Participants were continued to receive niraparib 200 mg and abiraterone acetate 1000 mg plus prednisone 10 mg in the open label extension phase.
- Cohort 1: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg: Participants with mCRPC and positive HRR gene alteration, received placebo in combination with abiraterone acetate 1000 mg tablet orally QD and prednisone 5 mg tablet orally BID (total dose 10 mg) in each 28 days treatment cycle starting from Cycle 1 Day 1 up to 29 months. Participants were then followed up for safety up to 5 years after last dose or until death, loss to follow-up, withdrawal of consent, or study termination. Participants who received placebo and abiraterone acetate plus prednisone were allowed to cross over to receive niraparib 200 mg and abiraterone acetate 1000 mg plus prednisone 10 mg in the open-label extension phase.
- Cohort 2: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg: Participants with mCRPC and negative HRR gene alteration, received niraparib 200 mg capsule in combination with abiraterone acetate 1000 mg tablet orally QD and prednisone 5 mg tablet orally BID (total dose 10 mg) in each 28 days treatment cycle starting from Cycle 1 Day 1 up to 29 months. Participants were then followed up for safety up to 5 years after last dose or until death, loss to follow-up, withdrawal of consent, or study termination. Participants were continued to receive niraparib 200 mg and abiraterone acetate 1000 mg plus prednisone 10 mg in the open label extension phase.
- Cohort 2: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg: Participants with mCRPC and negative HRR gene alteration, received placebo in combination with abiraterone acetate 1000 mg tablet orally QD and prednisone 5 mg tablet orally BID (total dose 10 mg) in each 28 days treatment cycle starting from Cycle 1 Day 1 up to 29 months. Participants were then followed up for safety up to 5 years after last dose or until death, loss to follow-up, withdrawal of consent, or study termination. Participants who received placebo and abiraterone acetate plus prednisone were allowed to cross over to receive niraparib 200 mg and abiraterone acetate 1000 mg plus prednisone 10 mg in the open-label extension phase.
- Cohort 3: Niraparib 200 mg and Abiraterone Acetate 1000 mg FDC + Prednisone 10 mg: Participants with mCRPC and positive HRR gene alteration, received fixed-dose combination (FDC) of niraparib 200 mg and abiraterone acetate 1000 mg combination tablet orally QD with prednisone 5 mg tablet orally BID (total dose 10 mg) in each 28 days treatment cycle starting from Cycle 1 Day 1 up to 9 months. Participants were then followed up for safety up to 5 years after last dose or until death, loss to follow-up, withdrawal of consent, or study termination. Participants were continued to receive same treatment in long-term extension phase.
Period: Overall Study
Arm/Group | Cohort 1: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 1: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 2: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 2: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 3: Niraparib 200 mg and Abiraterone Acetate 1000 mg FDC + Prednisone 10 mg
Started | 212 | 211 | 123 | 124 | 95
Breast Cancer Gene (BRCA) Subgroup | 113 | 112 | 0 | 0 | 52
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 212 | 211 | 123 | 124 | 95
Not completed — Ongoing | 155 | 148 | 66 | 79 | 84
Not completed — Death | 54 | 59 | 51 | 42 | 9
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 5 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 1: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 2: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 2: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 3: Niraparib 200 mg and Abiraterone Acetate 1000 mg FDC + Prednisone 10 mg | Total
Number analyzed (Participants) | 212 | 211 | 123 | 124 | 95 | 765
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (8.79) | 68.6 (8.17) | 71.2 (7.11) | 71.1 (7.52) | 69.2 (8.99) | 69.7 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 212 | 211 | 123 | 124 | 95 | 765
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 25 | 8 | 12 | 12 | 83
  Not Hispanic or Latino | 166 | 169 | 110 | 105 | 77 | 627
  Unknown or Not Reported | 20 | 17 | 5 | 7 | 6 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 1 | 3
  Asian | 29 | 41 | 45 | 37 | 14 | 166
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 5 | 0 | 0 | 0 | 3 | 8
  White | 160 | 153 | 72 | 83 | 70 | 538
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 17 | 16 | 5 | 4 | 7 | 49
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 2 | 5 | 2 | 7 | 2 | 18
  AUSTRALIA | 15 | 12 | 12 | 9 | 3 | 51
  BELGIUM | 5 | 1 | 2 | 3 | 0 | 11
  BRAZIL | 20 | 14 | 0 | 0 | 10 | 44
  BULGARIA | 1 | 0 | 0 | 0 | 0 | 1
  CANADA | 4 | 7 | 1 | 4 | 3 | 19
  CHINA | 7 | 4 | 0 | 0 | 0 | 11
  CZECH REPUBLIC | 4 | 3 | 1 | 2 | 1 | 11
  FRANCE | 13 | 12 | 5 | 4 | 3 | 37
  GERMANY | 0 | 4 | 0 | 0 | 5 | 9
  HUNGARY | 7 | 4 | 3 | 2 | 1 | 17
  ISRAEL | 0 | 0 | 0 | 0 | 3 | 3
  ITALY | 9 | 10 | 3 | 3 | 11 | 36
  MALAYSIA | 5 | 10 | 17 | 7 | 1 | 40
  MEXICO | 3 | 2 | 0 | 0 | 0 | 5
  NETHERLANDS | 3 | 4 | 2 | 2 | 0 | 11
  POLAND | 12 | 12 | 11 | 15 | 4 | 54
  PORTUGAL | 1 | 1 | 0 | 0 | 3 | 5
  RUSSIAN FEDERATION | 19 | 21 | 6 | 1 | 3 | 50
  SOUTH KOREA | 8 | 22 | 21 | 17 | 10 | 78
  SPAIN | 12 | 9 | 9 | 12 | 3 | 45
  SWEDEN | 4 | 2 | 1 | 1 | 1 | 9
  TAIWAN | 8 | 4 | 7 | 12 | 3 | 34
  TURKEY | 18 | 16 | 6 | 6 | 5 | 51
  UKRAINE | 18 | 20 | 12 | 11 | 9 | 70
  UNITED KINGDOM | 2 | 1 | 0 | 3 | 3 | 9
  UNITED STATES | 12 | 11 | 2 | 3 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Radiographic Progression-Free Survival (rPFS) as Assessed by Blinded Independent Central Review (BICR)
Description: As per BICR, rPFS is time interval from the date of randomization to radiographic progression or death, whichever occurred first. Radiographic progression was determined by: (1) progression of soft tissue lesions measured by computerized tomography (CT) or magnetic resonance imaging (MRI) as per response evaluation criteria in solid tumors (RECIST) 1.1; (2) Progression of bone lesions observed by bone scan based on prostate cancer working group 3 (PCWG3) criteria. PCWG3 criteria: bone progression was confirmed by subsequent scan greater than or equal to (>=) 6 weeks later. Week 8 scan was baseline to which all subsequent scans were compared to determine progression. Confirmatory scan >=2 new lesions indicate progression; scan does not show >=2 new lesions means no progression. If Week 8 scan less than (<) 2 new bone lesions compared to baseline, the initial scan >=2 new lesions compared to Week 8 scan indicates progression if confirmed by subsequent scan >=6 weeks later.
Time Frame: Up to 32 months
Population: The randomized analysis set for cohort 1 included all randomized participants in Cohort 1. Data for this outcome measure was planned to be collected and analyzed for Cohort 1 only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 1: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg
Number analyzed (Participants) | 212 | 211
Months | 16.46 [13.83 to 19.38] | 13.70 [10.91 to 16.39]
Statistical Analysis 1: Comparison: Cohort 1: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg vs Cohort 1: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg; Test type: Superiority; p = 0.0217, Log Rank; Hazard Ratio (HR) = 0.729, 95% CI 2-sided [0.556 to 0.956]

2. Primary Outcome: Cohort 1 Breast Cancer Gene (BRCA) Subgroup: Radiographic Progression-Free Survival (rPFS) as Assessed by Blinded Independent Central Review (BICR)
Description: As per BICR, rPFS is time interval from the date of randomization to radiographic progression or death, whichever occurred first. Radiographic progression was determined by: (1) progression of soft tissue lesions measured by CT or MRI as per RECIST 1.1; (2) Progression of bone lesions observed by bone scan based on PCWG3 criteria. PCWG3 criteria: bone progression was confirmed by subsequent scan >=6 weeks later. Week 8 scan was baseline to which all subsequent scans were compared to determine progression. Confirmatory scan >=2 new lesions indicate progression; scan does not show >=2 new lesions means no progression. If Week 8 scan <2 new bone lesions compared to baseline, the initial scan >=2 new lesions compared to Week 8 scan indicates progression if confirmed by subsequent scan >=6 weeks later.
Time Frame: Up to 32 months
Population: The randomized analysis set for cohort 1 BRCA subgroup included all randomized participants in Cohort 1 BRCA subgroup. Data for this outcome measure was planned to be collected and analyzed for BRCA subgroup of Cohort 1 only.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort 1 BRCA Subgroup: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg: Participants with metastatic castration-resistant prostate cancer (mCRPC) and BRCA alterations, received niraparib 200 milligrams (mg) capsule in combination with abiraterone acetate 1000 mg tablet orally once daily (QD) and prednisone 5 mg tablet orally twice daily (BID) (total dose 10 mg) in each 28 days treatment cycle starting from Cycle 1 Day 1 up to 29 months. Participants were then followed up for safety up to 5 years after last dose or until death, loss to follow-up, withdrawal of consent, or study termination. Participants were continued to receive niraparib 200 mg and abiraterone acetate 1000 mg plus prednisone 10 mg in the open label extension phase.
- Cohort 1 BRCA Subgroup: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg: Participants with mCRPC and BRCA alterations, received placebo in combination with abiraterone acetate 1000 mg tablet orally QD and prednisone 5 mg tablet orally BID (total dose 10 mg) in each 28 days treatment cycle starting from Cycle 1 Day 1 up to 29 months. Participants were then followed up for safety up to 5 years after last dose or until death, loss to follow-up, withdrawal of consent, or study termination. Participants who received placebo and abiraterone acetate plus prednisone were allowed to cross over to receive niraparib 200 mg and abiraterone acetate 1000 mg plus prednisone 10 mg in the open-label extension phase.
Arm/Group | Cohort 1 BRCA Subgroup: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 1 BRCA Subgroup: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg
Number analyzed (Participants) | 113 | 112
Months | 16.56 [13.86 to NA] — Here, NA signifies that upper limit of 95% confidence interval could not be calculated due to the too low number of participants with a rPFS event observed by the time of analysis. | 10.87 [8.31 to 13.80]
Statistical Analysis 1: Comparison: Cohort 1 BRCA Subgroup: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg vs Cohort 1 BRCA Subgroup: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg; Test type: Superiority; p = 0.0014, Log Rank; Hazard Ratio (HR) = 0.533, 95% CI 2-sided [0.361 to 0.789]

3. Secondary Outcome: Cohort 1: Overall Survival (OS)
Time Frame: Up to 97 months
Reporting Status: Not Posted, anticipated posting 2028-02

4. Secondary Outcome: Cohort 1: Time to Symptomatic Progression
Time Frame: Up to 97 months
Reporting Status: Not Posted, anticipated posting 2028-02

5. Secondary Outcome: Cohort 1: Time to Initiation of Cytotoxic Chemotherapy
Time Frame: Up to 97 months
Reporting Status: Not Posted, anticipated posting 2028-02

6. Secondary Outcome: Observed Plasma Concentrations of Niraparib
Time Frame: Up to 97 months
Reporting Status: Not Posted, anticipated posting 2028-02

7. Secondary Outcome: Observed Plasma Concentrations of Abiraterone
Time Frame: Up to 97 months
Reporting Status: Not Posted, anticipated posting 2028-02

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Time Frame: Up to 96 months
Reporting Status: Not Posted, anticipated posting 2028-02

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events by Severity
Time Frame: Up to 96 months
Reporting Status: Not Posted, anticipated posting 2028-02

10. Secondary Outcome: Number of Participants With Abnormalities in Laboratory Values
Time Frame: Up to 96 months
Reporting Status: Not Posted, anticipated posting 2028-02

ADVERSE EVENTS:
Time Frame: Up to 32 months
Description: The safety analysis set for Cohort 1 and Cohort 2 included all randomized participants who received at least 1 dose of study drug in Cohort 1 or Cohort 2. The safety analysis set for Cohort 3 included all participants who received at least 1 dose of study drug in Cohort 3.
Arm/Group | Cohort 1: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 1: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 2: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 2: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg | Cohort 3: Niraparib 200 mg and Abiraterone Acetate 1000 mg FDC + Prednisone 10 mg
All-Cause Mortality (participants affected / at risk) | 55/212 | 59/211 | 53/123 | 44/123 | 9/95
Serious Adverse Events (participants affected / at risk) | 76/212 | 52/211 | 66/123 | 45/123 | 21/95
Other Adverse Events (participants affected / at risk) | 198/212 | 178/211 | 117/123 | 108/123 | 83/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg (N=212) | Cohort 1: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg (N=211) | Cohort 2: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg (N=123) | Cohort 2: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg (N=123) | Cohort 3: Niraparib 200 mg and Abiraterone Acetate 1000 mg FDC + Prednisone 10 mg (N=95)
Anaemia (Blood and lymphatic system disorders) | 12 | 2 | 20 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphoid Tissue Hyperplasia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 2 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Arrhythmia Supraventricular (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1 | 2 | 0
Cardiac Failure (Cardiac disorders) | 1 | 1 | 3 | 0 | 0
Cardiac Failure Acute (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cor Pulmonale (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 2 | 0 | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 3 | 3 | 0 | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Blindness Unilateral (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye Pain (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Adverse Drug Reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 2 | 1 | 0
Gait Disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 1 | 1 | 0 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 0 | 2 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatitis Acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Abscess Oral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 6 | 1 | 3 | 0 | 0
Covid-19 Pneumonia (Infections and infestations) | 4 | 2 | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Medical Device Site Joint Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Meningitis Aseptic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 4 | 4 | 2 | 2
Post Procedural Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Suspected Covid-19 (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 2 | 2 | 1 | 2
Urosepsis (Infections and infestations) | 2 | 1 | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cardiac Valve Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post Procedural Pulmonary Embolism (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Radiation Proctitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Vaccination Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung Adenocarcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cauda Equina Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral Arteriosclerosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Depressed Level of Consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Malignant Spinal Cord Compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Peroneal Nerve Palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Vascular Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 2 | 3 | 1 | 1
Bladder Mass (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Bladder Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Bladder Perforation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Calculus Bladder (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 3 | 1 | 2 | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0
Micturition Disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 4 | 2 | 0 | 3 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 2 | 3
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Circulatory Collapse (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypovolaemic Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Iliac Artery Rupture (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 1 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg (N=212) | Cohort 1: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg (N=211) | Cohort 2: Niraparib 200 mg + Abiraterone Acetate 1000 mg + Prednisone 10 mg (N=123) | Cohort 2: Placebo + Abiraterone Acetate 1000 mg + Prednisone 10 mg (N=123) | Cohort 3: Niraparib 200 mg and Abiraterone Acetate 1000 mg FDC + Prednisone 10 mg (N=95)
Anaemia (Blood and lymphatic system disorders) | 95 | 43 | 59 | 19 | 37
Leukopenia (Blood and lymphatic system disorders) | 22 | 5 | 7 | 2 | 3
Lymphopenia (Blood and lymphatic system disorders) | 19 | 4 | 8 | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 28 | 12 | 21 | 6 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 45 | 18 | 24 | 3 | 11
Abdominal Distension (Gastrointestinal disorders) | 8 | 1 | 5 | 2 | 7
Abdominal Pain (Gastrointestinal disorders) | 9 | 12 | 2 | 4 | 2
Constipation (Gastrointestinal disorders) | 65 | 29 | 38 | 25 | 23
Diarrhoea (Gastrointestinal disorders) | 10 | 8 | 10 | 9 | 5
Dry Mouth (Gastrointestinal disorders) | 6 | 3 | 5 | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 13 | 6 | 8 | 7 | 6
Gastritis (Gastrointestinal disorders) | 3 | 3 | 7 | 4 | 2
Nausea (Gastrointestinal disorders) | 50 | 29 | 29 | 20 | 25
Vomiting (Gastrointestinal disorders) | 28 | 14 | 17 | 11 | 8
Asthenia (General disorders) | 33 | 19 | 22 | 14 | 12
Fatigue (General disorders) | 56 | 35 | 29 | 21 | 16
Oedema Peripheral (General disorders) | 20 | 18 | 16 | 15 | 0
Pyrexia (General disorders) | 12 | 11 | 6 | 3 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 8 | 7 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 19 | 11 | 9 | 5 | 3
Fall (Injury, poisoning and procedural complications) | 11 | 25 | 9 | 16 | 4
Alanine Aminotransferase Increased (Investigations) | 10 | 22 | 7 | 11 | 2
Aspartate Aminotransferase Increased (Investigations) | 11 | 20 | 6 | 12 | 4
Blood Alkaline Phosphatase Increased (Investigations) | 21 | 14 | 9 | 7 | 5
Blood Creatinine Increased (Investigations) | 19 | 8 | 5 | 3 | 7
Weight Decreased (Investigations) | 19 | 5 | 20 | 8 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 30 | 13 | 29 | 11 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 21 | 18 | 18 | 10 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 18 | 12 | 9 | 6 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 27 | 19 | 15 | 9 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 5 | 2 | 0 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 20 | 11 | 20 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 31 | 44 | 19 | 25 | 7
Bone Pain (Musculoskeletal and connective tissue disorders) | 21 | 24 | 10 | 8 | 5
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 7 | 4 | 9 | 9 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 | 11 | 4 | 7 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 10 | 14 | 9 | 13 | 4
Dizziness (Nervous system disorders) | 24 | 12 | 13 | 13 | 2
Headache (Nervous system disorders) | 16 | 19 | 3 | 6 | 7
Insomnia (Psychiatric disorders) | 22 | 8 | 8 | 7 | 3
Haematuria (Renal and urinary disorders) | 12 | 8 | 7 | 9 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 10 | 6 | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 12 | 15 | 8 | 6
Hot Flush (Vascular disorders) | 15 | 15 | 6 | 13 | 4
Hypertension (Vascular disorders) | 66 | 44 | 41 | 27 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03748641/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT03748641/SAP_001.pdf